CLINICAL TRIAL: NCT00931762
Title: Phase II Trial of Oral Panobinostat (LBH589), a Novel Deacetylase Inhibitor (DACi) in Patients With Primary Myelofibrosis (PMF), Post Essential Thrombocythemia (ET) Myelofibrosis and Post- Polycythemia Vera (PV) Myelofibrosis
Brief Title: A Study to Evaluate Safety and Efficacy of Panobinostat in Participants With Primary Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BUS58
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera; Post-Essential Thrombocytopenia
Keywords: Bone marrow; Myelofibrosis; JAK2mutation; Post-Polycythemia Vera; Post-Essential Thrombocytopenia
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (Experimental): Participants received panobinostat 40 mg, capsules, orally, with or without food, three times a week on Monday, Wednesday, and Friday for up to 6 treatment cycles (each cycle of 28-days) with dose adjustments possible.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat oral capsules
  Other Names: LBH589; H-DAC Inhibitor

SUMMARY:
This study assessed the safety and efficacy of Panobinostat as a single agent in the treatment of Primary Myelofibrosis, Post-Polycythemia Vera and Post-Essential Thrombocythemia. There were two cohorts - participants with JAK2 mutation and participants without JAK2 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of myelofibrosis, either primary myelofibrosis (PMF), post- polycythemia vera (PV) or post-essential thrombocythemia (ET) myelofibrosis (MF) with international prognostic scoring system (IPSS) score of 2 (intermediate risk) or 3 (high risk) plus at least one of the following:

   Symptomatic spenomegaly (≥10 centimeter [cm] below costal margin [BCM]) Hemoglobin < 10 or red cell transfusion dependent. (The presence of a janus kinase (JAK2) V617F mutation is not required for study entry).
2. Participants must meet the following laboratory criteria:

   * Participants can be either JAK2 V617F mutated or wild type.
   * Serum potassium, magnesium, phosphorous, sodium, total calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL) for the institution Note: Potassium, magnesium, phosphorous, sodium, and/or calcium supplements maybe given to correct values that are < lower limit of normal (LLN). Post correction values must not be deemed to be a clinically significant abnormality prior to participants being dosed.
   * Creatinine < 1.5 X upper limit of normal (ULN) or calculated creatinine clearance (CrCl) ≥ 50 milliliter per minute (mL/min) (modification of diet in renal diseases [MDRD] formula).
   * Aspartate aminotransferase [AST] and alanine transaminase [ALT] ≤ 2.5 x ULN.
   * Serum total bilirubin ≤ 1.5 x ULN.
3. Eastern cooperative oncology group (ECOG) performance status of ≤ 2.
4. Clinically euthyroid. Note: Participants are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.

Exclusion Criteria:

1. Prior histone deacetylases (HDAC), deacetylase (DAC), heat shock protein 90 (HSP90) inhibitors or valproic acid for the treatment of cancer.
2. Previous treatment with JAK2 inhibitors.
3. Any participant who has previously received radiation therapy to ≥ 30% of the bone marrow.
4. Impaired cardiac function or clinically significant cardiac diseases.
5. Participant with unresolved diarrhoea ≥ grade 2.
6. Participants using medications that have a relative risk of prolonging the QT interval or inducing Torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug.
7. Participants who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of surgery.
8. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test at screening and at baseline.
9. Male participants whose sexual partners are WOCBP not using effective birth control.
10. Participants with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix).
11. Participants with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2011-08-29 (Actual); Study Completion 2011-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (9):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - New York Presbyterian Hospital - Weill Cornell Medical College, New York, New York

REFERENCES:
- [Result] DeAngelo DJ, Mesa RA, Fiskus W, Tefferi A, Paley C, Wadleigh M, Ritchie EK, Snyder DS, Begna K, Ganguly S, Ondovik MS, Rine J, Bhalla KN. Phase II trial of panobinostat, an oral pan-deacetylase inhibitor in patients with primary myelofibrosis, post-essential thrombocythaemia, and post-polycythaemia vera myelofibrosis. Br J Haematol. 2013 Aug;162(3):326-35. doi: 10.1111/bjh.12384. Epub 2013 May 23. PMID 23701016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 investigative centers in the United States from 31 August 2009 to 29 August 2011.
Period: Overall Study
Arm/Group | Panobinostat
Started | 35
Completed | 0
Not Completed | 35
Not completed — Abnormal Laboratory Value (s) | 2
Not completed — Administrative Problems | 5
Not completed — Death | 1
Not completed — Disease Progression | 3
Not completed — Adverse Event (s) | 11
Not completed — Subject withdrew consent | 13

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) population included all participants who received at least one dose of study drug.
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Rate Per International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) Criteria
Description: Overall response (OR) = Complete remission (CR) + Partial remission (PR) + Clinical improvement (CI). CR: complete resolution of disease-related symptoms and signs with hemoglobin level 110 grams per deciliter (g/L), platelet count 100 x 10^9/liter (L), and absolute neutrophil count (ANC) 1.0 x 10^9/L, all 3 blood counts < upper normal limit (UNL), normal leukocyte differential, and bone marrow histologic remission. PR= all of the criteria for CR except the requirement for bone marrow histologic remission. CI= minimum 20 g/L increase in hemoglobin for transfusion or becoming transfusion independent or reduction in splenomegaly ≥ 50% or 100% increase in platelet count and absolute platelet count of 50 x 10^9/L and 100% increase in ANC of at least 0.5 x 10^9/L.
Time Frame: Up to approximately 2 years
Population: FAS population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
percentage of participants | 2.9 [0.1 to 14.9]

2. Secondary Outcome: Change From Baseline in Myelofibrosis Symptom Assessment Form (MF-SAF) Scale Scores At Cycle 6
Description: The MF-SAF consists of seven questions about key symptoms and impact of MF. Questions were scored on a scale of 0-10, with higher scores indicating more severe symptoms and greater inactivity. Questions 1-6 investigate the following symptoms: night sweats, pruritus/itching, abdominal discomfort, pain under the ribs, early satiety and bone/muscle pain. Question 7 asked participants to report levels of inactivity. Negative change from baseline indicates improvement.
Time Frame: Baseline, Cycle 6 (each cycle was of 28 days)
Population: FAS population included all participants who received at least one dose of study drug.
  All 35 participants were evaluated for this Outcome. The Number Analyzed represented in each row differs from the Overall Number of Participants Analyzed as scores that are presented are for the participants who reported the measured event at the time evaluated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
score on a scale
  Cycle 6, Day 1: Fatigue Right now: number analyzed (Participants) | 2
  Cycle 6, Day 1: Fatigue Right now | -1.5 (2.12)
  Cycle 6, Day 1: Fatigue Usual Past 24 Hours: number analyzed (Participants) | 2
  Cycle 6, Day 1: Fatigue Usual Past 24 Hours | -1.0 (5.66)
  Cycle 6, Day 1: Fatigue Worst Past 24 Hours: number analyzed (Participants) | 2
  Cycle 6, Day 1: Fatigue Worst Past 24 Hours | -3.0 (2.83)
  Cycle 6, Day 1: General Activity: number analyzed (Participants) | 2
  Cycle 6, Day 1: General Activity | -3.5 (2.12)
  Cycle 6, Day 1: Mood: number analyzed (Participants) | 2
  Cycle 6, Day 1: Mood | -3.5 (3.54)
  Cycle 6, Day 1: Walking Ability: number analyzed (Participants) | 2
  Cycle 6, Day 1: Walking Ability | -3.0 (5.66)
  Cycle 6, Day 1: Normal Work: number analyzed (Participants) | 2
  Cycle 6, Day 1: Normal Work | -4.0 (4.24)
  Cycle 6, Day 1: Relations with Other People: number analyzed (Participants) | 2
  Cycle 6, Day 1: Relations with Other People | -4.5 (2.12)
  Cycle 6, Day 1: Enjoyment of Life: number analyzed (Participants) | 2
  Cycle 6, Day 1: Enjoyment of Life | -5.0 (4.24)
  Cycle 6, Day 1: Filling up quickly when you eat: number analyzed (Participants) | 2
  Cycle 6, Day 1: Filling up quickly when you eat | 1.0 (1.41)
  Cycle 6, Day 1: Abdominal pain or Discomfort: number analyzed (Participants) | 2
  Cycle 6, Day 1: Abdominal pain or Discomfort | 0.5 (2.12)
  Cycle 6, Day 1: Inactivity: number analyzed (Participants) | 2
  Cycle 6, Day 1: Inactivity | -0.5 (3.54)
  Cycle 6, Day 1: Cough: number analyzed (Participants) | 2
  Cycle 6, Day 1: Cough | -1.5 (2.12)
  Cycle 6, Day 1: Night Sweats: number analyzed (Participants) | 2
  Cycle 6, Day 1: Night Sweats | -0.5 (0.71)
  Cycle 6, Day 1: Itching: number analyzed (Participants) | 2
  Cycle 6, Day 1: Itching | 1.5 (2.12)
  Cycle 6, Day 1: Bone Pain: number analyzed (Participants) | 2
  Cycle 6, Day 1: Bone Pain | -2.5 (0.71)
  Cycle 6, Day 1: What is Overall Quality of Life?: number analyzed (Participants) | 2
  Cycle 6, Day 1: What is Overall Quality of Life? | -2.5 (2.12)

3. Secondary Outcome: Change From Baseline in Myelofibrosis Symptom Assessment Form (MF-SAF) Scale Scores
Description: as for outcome 2
Time Frame: Baseline, Cycles 2, and 4 (each cycle was of 28-days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
score on a scale
  Cycle 2, Day 1: Fatigue Right now: number analyzed (Participants) | 23
  Cycle 2, Day 1: Fatigue Right now | 0.0 (2.00)
  Cycle 2, Day 1: Fatigue Usual Past 24 Hours: number analyzed (Participants) | 23
  Cycle 2, Day 1: Fatigue Usual Past 24 Hours | 0.5 (1.83)
  Cycle 2, Day 1: Fatigue Worst Past 24 Hours: number analyzed (Participants) | 23
  Cycle 2, Day 1: Fatigue Worst Past 24 Hours | 0.7 (1.98)
  Cycle 2, Day 1: General Activity: number analyzed (Participants) | 23
  Cycle 2, Day 1: General Activity | 0.0 (2.03)
  Cycle 2, Day 1: Mood: number analyzed (Participants) | 22
  Cycle 2, Day 1: Mood | 0.5 (2.15)
  Cycle 2, Day 1: Walking Ability: number analyzed (Participants) | 23
  Cycle 2, Day 1: Walking Ability | -0.6 (2.86)
  Cycle 2, Day 1: Normal Work: number analyzed (Participants) | 23
  Cycle 2, Day 1: Normal Work | 0.2 (2.87)
  Cycle 2, Day 1: Relations with Other People: number analyzed (Participants) | 23
  Cycle 2, Day 1: Relations with Other People | -0.1 (2.71)
  Cycle 2, Day 1: Enjoyment of Life: number analyzed (Participants) | 23
  Cycle 2, Day 1: Enjoyment of Life | 0.3 (3.30)
  Cycle 2, Day 1: Filling up quickly when you eat: number analyzed (Participants) | 23
  Cycle 2, Day 1: Filling up quickly when you eat | 0.7 (2.38)
  Cycle 2, Day 1: Abdominal Pain or Discomfort: number analyzed (Participants) | 23
  Cycle 2, Day 1: Abdominal Pain or Discomfort | -0.0 (2.64)
  Cycle 2, Day 1: Inactivity: number analyzed (Participants) | 23
  Cycle 2, Day 1: Inactivity | 0.8 (2.45)
  Cycle 2, Day 1: Cough: number analyzed (Participants) | 22
  Cycle 2, Day 1: Cough | -0.1 (2.07)
  Cycle 2, Day 1: Night Sweats: number analyzed (Participants) | 23
  Cycle 2, Day 1: Night Sweats | -1.0 (2.36)
  Cycle 2, Day 1: Itching: number analyzed (Participants) | 21
  Cycle 2, Day 1: Itching | -1.5 (2.89)
  Cycle 2, Day 1: Bone Pain: number analyzed (Participants) | 22
  Cycle 2, Day 1: Bone Pain | -1.0 (2.79)
  Cycle 2, Day 1: What is Overall Quality of Life?: number analyzed (Participants) | 22
  Cycle 2, Day 1: What is Overall Quality of Life? | -0.4 (2.24)
  Cycle 4, Day 1: Fatigue Right now: number analyzed (Participants) | 8
  Cycle 4, Day 1: Fatigue Right now | 0.0 (1.93)
  Cycle 4, Day 1: Fatigue Usual Past 24 Hours: number analyzed (Participants) | 8
  Cycle 4, Day 1: Fatigue Usual Past 24 Hours | 0.8 (1.91)
  Cycle 4, Day 1: Fatigue Worst Past 24 Hours: number analyzed (Participants) | 8
  Cycle 4, Day 1: Fatigue Worst Past 24 Hours | 1.0 (1.31)
  Cycle 4, Day 1: General Activity: number analyzed (Participants) | 8
  Cycle 4, Day 1: General Activity | -0.5 (3.07)
  Cycle 4, Day 1: Mood: number analyzed (Participants) | 7
  Cycle 4, Day 1: Mood | 0.3 (2.75)
  Cycle 4, Day 1: Walking Ability: number analyzed (Participants) | 7
  Cycle 4, Day 1: Walking Ability | -0.6 (3.26)
  Cycle 4, Day 1: Normal Work: number analyzed (Participants) | 8
  Cycle 4, Day 1: Normal Work | 0.9 (2.53)
  Cycle 4, Day 1: Relations with Other People: number analyzed (Participants) | 8
  Cycle 4, Day 1: Relations with Other People | -0.6 (2.20)
  Cycle 4, Day 1: Enjoyment of Life: number analyzed (Participants) | 8
  Cycle 4, Day 1: Enjoyment of Life | 0.4 (3.62)
  Cycle 4, Day 1: Filling up quickly when you eat: number analyzed (Participants) | 8
  Cycle 4, Day 1: Filling up quickly when you eat | -0.1 (4.42)
  Cycle 4, Day 1: Abdominal Pain or Discomfort: number analyzed (Participants) | 8
  Cycle 4, Day 1: Abdominal Pain or Discomfort | 1.0 (2.67)
  Cycle 4, Day 1: Inactivity: number analyzed (Participants) | 8
  Cycle 4, Day 1: Inactivity | 0.6 (3.25)
  Cycle 4, Day 1: Cough: number analyzed (Participants) | 8
  Cycle 4, Day 1: Cough | -0.9 (1.36)
  Cycle 4, Day 1: Night Sweats: number analyzed (Participants) | 8
  Cycle 4, Day 1: Night Sweats | -1.1 (3.52)
  Cycle 4, Day 1: Itching: number analyzed (Participants) | 7
  Cycle 4, Day 1: Itching | -0.1 (0.90)
  Cycle 4, Day 1: Bone Pain: number analyzed (Participants) | 8
  Cycle 4, Day 1: Bone Pain | -1.8 (3.41)
  Cycle 4, Day 1: What is Overall Quality of Life?: number analyzed (Participants) | 7
  Cycle 4, Day 1: What is Overall Quality of Life? | -0.3 (1.60)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs), and Serious Adverse Events (SAEs)
Description: An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. SAEs was an undesirable sign, symptom or medical condition which is: life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, requires hospitalizations or prolongation of hospitalizations, or is medically significant
Time Frame: AE: From the start of treatment up to 28 days after last study dose (up to approximately 2 years); SAE: From time of informed consent up to 4 weeks after last study dose (approximately 2 years)
Population: Safety set population included all participants who received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
Participants
  AEs | 35
  SAEs | 19

5. Other Pre Specified Outcome: Monthly Capsule Counts to Assess Compliance to Panobinostat Treatment
Time Frame: Up to approximately 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: To Compare the Response to Panobinostat in Patients With the JAK2 V617F Mutation to Those Without the JAK2 V617F Mutation
Time Frame: Up to approximately 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE: From the start of treatment up to 28 days after last study dose (up to approximately 2 years); SAE: From time of informed consent up to 4 weeks after last study dose (approximately 2 years)
Description: Safety set population included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Panobinostat
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 19/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=35)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Haemoglobin decreased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=35)
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Cushingoid (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Eye haemorrhage (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 19
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 4
Chills (General disorders) | 4
Fatigue (General disorders) | 20
Feeling jittery (General disorders) | 1
General physical health deterioration (General disorders) | 1
Generalised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 2
Pyrexia (General disorders) | 6
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Candidiasis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 4
Blood magnesium decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
International normalised ratio increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.